CLINICAL TRIAL: NCT03049020
Title: The Efficacy of Laparoscopic Sacrocolpopexy in the Treatment of Pelvic Organ Prolapse in Women With or Without Avulsion of the Levator Ani Muscle
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Kamil Svabik, Kamil Svabik, MD, Ph.D., Charles University, Czech Republic
Other Study IDs: 1760/14S-IV
Record Dates: First submitted 2015-12-10; First posted 2017-02-09 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Pelvic Organ Prolapse Recurrence
Keywords: pelvic organ prolapse; sacrocolpopexy; pelvic floor ultrasound
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- With levator ani avulsion: Patients indicated for sacrocolpopexy for pelvic organ prolapse and suffering with levator ani avulsion
  Interventions: Procedure: laparoscopic sacrocolpopexy
- Without levator ani avulsion: Patients indicated for sacrocolpopexy for pelvic organ prolapse and without levator ani avulsion
  Interventions: Procedure: laparoscopic sacrocolpopexy

INTERVENTIONS:
Procedure: laparoscopic sacrocolpopexy — standard laparoscopic sacrocolpopexy for prolapse treatment

SUMMARY:
Based on a prospective study, to evaluate how pre-operative pelvic floor status - the presence of injury to the musculus levator ani - may influence the results of laparoscopic sacrocolpopexy. The investigators hope to confirm or disprove the hypothesis that the presence of such injury increases the risk of post-operative prolapse recurrence

DETAILED DESCRIPTION:
Introduction Pelvic organ prolapse (POP), is a common health problem affecting up to 40% of women. The life time risk for undergoing at least one session of pelvic organ prolapse surgery has been estimated at approximately 13%. The prevalence of reoperation after primary pelvic reconstructive surgery is high, around 30%, while some articles report the figure as up to 58%. From the beginning of the 1990s the view of pelvic floor defects and urinary incontinence in women started to change significantly. The diagnostics and management of these defects became an independent uro-gynecological sub-specialization within gynecology and obstetrics, and it has been included among 4 basic sub-specializations recognized by the European Board and College of Obstetrics and Gynecology. Surgical treatment is indicated in women with symptomatic POP when conservative management has failed or has been declined. There is no indication for repair of asymptomatic POP as an isolated procedure where surgical correction is of uncertain benefit and adds peri- and post-operative risks. The objective of our treatment should always aim to restore quality of life and comfort. Very little is known of the factors associated with surgical failure. Studies have identified a variety of risk factors: younger age, high body mass index and advanced preoperative prolapse (grade III-IV) were associated with an increased risk of reoperation in some studies, while other studies did not prove these hypotheses. One factor which significantly influences the result of the pelvic organ surgery is the presence of pelvic floor injury. Injury of the levator ani muscle mainly affects the results of traditional vaginal wall repair, with 60% risk of recurrence. In the last few years, in an attempt to reduce recurrence and improve the outcome of reconstructive surgery in the treatment of pelvic organ prolapse, surgeons have started to use transvaginally introduced prosthetic material (mesh). This type of surgery significantly increases the efficacy of the procedure (anatomic cure rate over 90%), but its use is associated with a risk of some complications (vaginal erosions and potential consecutive infections, granulomas, dyspareunia, vesico-vaginal fistulas, chronic pain) thereby potentially reducing the patients' quality of life and leading to additional surgery. If the mesh is introduced during the sacrocolpopexy and the vaginal wall is not open, there is a significant decrease of mesh-related complications. Laparoscopic sacrocolpopexy is considered the gold standard for the management of apical prolapse with high long-term efficacy. Based on the retrospective data available, it seems that the status of the pelvic floor may also influence the results of this procedure, but at present investigators have no data to confirm this hypothesis. Therefore investigators plan to obtain these data from a prospective analysis of the results of laparoscopic sacrocolpopexy.

For the prospective longitudinal study, the investigators plan to include all patients for whom surgical treatment of pelvic organ prolapse and laparoscopic sacrocolpopexy are indicated. Based on pre-study power analysis enrollment of 120 patients is planned (after preliminary evaluation of the results this could be increased to 160 patients), which is the minimal number to prove or disprove the null hypothesis: The pelvic floor does not influence the result of laparoscopic sacrocolpopexy in women with symptomatic pelvic organ prolapse stage II or higher. Based on previous studies it can be anticipated that the failure rate in patients with a defect of the pelvic floor will be higher. To enroll an adequate number of patients the study will be conducted in two university centers with long experience of this type of surgery (the number of enrolled patients in each workplace should be identical). Based on pre-study statistical calculations (power analysis) it is indicated that the required sample size for final statistical analysis in each group is 54 patients (allocation ratio 1:1). Investigators estimate a drop-out rate of 10%, therefore it is planned to enroll 60 patients into each group.

Aim of the study Based on a prospective study, to evaluate how pre-operative pelvic floor status - the presence of injury to the musculus levator ani - may influence the results of laparoscopic sacrocolpopexy. The investigators hope to confirm or disprove the hypothesis that the presence of such injury increases the risk of post-operative prolapse recurrence.

Inclusion criteria are:

Age over 18, signed informed consent, symptomatic pelvic organ prolapse stage II or higher (according to the International Continence Society Pelvic Organ Prolapse quantification system - POPQ) in anterior and apical (central) compartment, and agreement with postoperative follow-up.

Exclusion criteria are:

Previous pelvic reconstructive surgery with mesh, isolated posterior compartment prolapse, previous radiotherapy in lesser pelvis, contraindication for laparoscopic sacrocolpopexy.

Pre-operative assessment.

All patients will undergo complete urogynecological investigation before the procedure: history, clinical examination, assessment of pelvic organ prolapse using the POPQ system, examination of the levator resting tone and contraction (Oxford scale),where appropriate urodynamics according to International Continence Society recommendation and ultrasound examination. They will also complete standardized international questionnaires (ICIQ-UI SF, PISQ 12, POPDI). Ultrasound examinations will be performed as a combined examination using a convex probe, from abdominal and perineal approaches, and sectoral vaginal probe from the introital approach. The study will be recorded mainly in digital form. Acquired data from 4D imagery will be preserved in form of data set and processed with the appropriate proper software. The ultrasound examination will include an assessment of standard parameters describing position of urethrovesical junction, bladder descent, uterus descent, posterior vaginal wall descent (rectocele, enterocele). Using 3D/4D ultrasound examination the status of pelvic floor will be evaluated (presence of avulsion of puborectalis muscle, abnormal genital hiatus distension). Based on pre-operative ultrasound examination, the women will be divided into two groups:

1. Group - women without defect of pelvic floor with urogenital hiatus size up to 30 cm2
2. Group - women with pelvic floor trauma with urogenital hiatus size over 30 cm2

Surgery and peri-operative monitoring All surgical procedures will be provided under general anesthesia, and antibiotic prophylaxis will be used. Surgery will be provided in standardized steps: identification of the promontory, dissection of the peritoneum above the promontory and preparation of the ligamentum longitudinale anterior, peritoneum dissection, dissection of the vesicovaginal septum up to bladder neck, dissection of the rectovaginal septum towards the perineum, application of Y mesh, fixation to the vaginal apex using the non-absorbable sutures, and for anterior and posterior vaginal wall absorbable sutures fixation of the upper mesh arm to the ligamentum longitudinale anterior using non-absorbable suture, following by complete peritoneum closure above the mesh. The procedure could include salpingo-oophorectomy, supracervical hysterectomy or total hysterectomy (concomitant procedures are not exclusion criteria).

Any peri-operative complications will be monitored. Surgical evaluation will include operating time (from incision to last suture), estimated intraoperative blood loss (vacuum aspiration), and perioperative complications (bladder perforation, vagina perforation, bowel injury, ureter injury and vascular injury). Postoperative data will be analyzed, including early postoperative complications (hematoma, spontaneous voiding recovery, urinary tract infection, ileus, constipation) and late postoperative complications (procedure failure, mesh erosion, de novo voiding difficulty, de novo stress urinary incontinence, further surgical procedures).

Post-operative follow-up The first post-operative complete examination is planned for 3 months after surgery (the same examination as before the procedure). The next check-up will be provided one year and two years after surgery, and the procedure will be the same as at the 3-month check-up. In addition to pre-operative ultrasound examination, the position of the mesh will be monitored. We plan to have a minimum one year follow-up for all patients in this study, and also after two years when possible. Postoperative follow-up will be terminated if the result of surgery is evaluated as a failure, and in these cases reoperation will be offered. We also plan further post-operative follow-up up to five years.

Criteria for evaluation of the cure and failure:

Primary outcome: the objective cure will be defined as absence of pelvic organ prolapse (using the POPQ system - maximal I. stage prolapse).

Number of failures in each group: failure is defined as pelvic organ prolapse stage II or higher using the POPQ system during the clinical examination, or as a descent 1 cm below the lower edge of the pubic bone based on ultrasound examination .

Secondary outcome:

These include change of the genital hiatus size, distance of mesh from the bladder neck urethrovesical junction), lowest position of the mesh, evaluation of the subjective parameters, quality of life based on evaluation of questionnaires ICIQ-SF, PISQ 12, POPDI, occurrence of de novo stress urinary incontinence, number of re-operations for pelvic organ prolapse, occurrence de novo symptoms of overactive bladder, in sexually active patients occurrence of de novo dyspareunia

Our project completely fulfills the primary aims in conception of health research till the year 2022, in the subfield "Innovative surgical procedure". Basic aims and priorities of the project are: implementation of the surgical procedures with lower invasivity to the treatment of pelvic organ prolapse and predict its efficacy on pre-operative pelvic floor status, minimizing unfavorable impact of the surgical procedure on the patient. Basis for the evaluation of the socio-economic contribution of the project solution will be high-quality evaluation of modern surgical procedures. Implementation of the new effective procedures for the pelvic organ prolapse shall significantly decrease total treatment cost, and significantly improve the long term quality of life of the patient. Thus is necessary to conduct such type of study, in order to use only those procedures which improve or maintain treatment effectiveness, do not increase the complication rate, and decrease the recovery time - thus having a fundamental impact on the amount of money invested from the public budget.

d) Methods promotion For a comparison of two groups of patient, with or without pelvic floor injury is estimated range selections in particular groups. If we mark p1 percentage of success rate procedure in patient with pelvic floor injury, p2 percentage of success rate procedure in the group without pelvic floor injury, for a 5% significance level we will prove zero hypothesis (that the percentage success rate is in all groups same) or the alternative hypothesis (that the percentage success rate differ). We require the ranges of selection to be the same in all groups same, and for percent values p1=85%, P2=60% a we require power test 80%. Under these conditions statistical calculations indicate that the required sample size in each group is 54 patients, and so as a whole we will analyze the data of almost 108 patients. We estimate a drop-out rate of 10%, so it is planned to enrolled 60 patients into each group- total 120 patients. The success rate used to calculate the size of the group has been estimated from previous studies; the estimated success rate of 60% for the patient with pelvic floor defect, and higher efficacy in patient with normal pelvic floor (85%). After evaluation of one year result of 60 women we plan to provide interim analysis and re-calculated the numbers of women which should be enrolled to the study to reach the statistical significance, and we are able to increase the number of enrolled women up to 20 in each center to total number of 160 included patients. Based on a statistical model, special software for data input will be prepared. The values to be monitored will be exactly specified in the model to allow for subsequent statistical processing. In our study we will use several types of statistical evaluation. In the tables summarizing general characteristics, data will be evaluated by means of data average and median, significant deviation. Furthermore, we will establish floor and cap of 95% confidence interval to arrive at an average. Zero or alternative hypotheses will be established and their validity determined. Where numbers are compared, chi square will be applied, while in cases where the number of observations is small, Fischer exact test will be used. We will be used non-parametric Kruskal-Wallis one-way analysis of variance for quantitative features and Fisher exact test for contingency tables. We used Bonferroni inequality to correct p value in case of multiple comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* signed informed consent
* symptomatic pelvic organ prolapse stage II or higher (according to the International Continence Society Pelvic Organ Prolapse quantification system - POPQ) in anterior and apical (central) compartment
* agreement with postoperative follow-up

Exclusion Criteria:

* Previous pelvic reconstructive mesh surgery
* Isolated posterior compartment prolapse
* Previous radiotherapy in lesser pelvis
* Contraindication of laparoscopic sacrocolpopexy

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age over 18, symptomatic pelvic organ prolapse stage II or higher (according to the International Continence Society Pelvic Organ Prolapse quantification system - POPQ) in anterior and apical (central) compartment
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Objective cure rate | One year
  The objective cure will be defined as absence of pelvic organ prolapse. Number of failures in each group: failure is defined as pelvic organ prolapse stage II or higher using the POPQ system during the clinical examination, or as a descent 1 cm below the lower edge of the pubic bone based on ultrasound examination

SECONDARY OUTCOMES:
Genital hiatus size | One year
  Evaluated on Valsalva in 4D transperineal ultrasound rendered volumes
Distance of mesh from the bladder neck | One year
  measured in sagittal plane on transperineal ultrasound.
Lowest position of the mesh | One year
  measured in sagittal plane on transperineal ultrasound.
ICIQ-UI SF | One year
  International Consultation on Incontinence Questionnaire - Urinary Incontinence , short form.
PISQ 12 | One year
  Pelvic Organ Prolapse/ Incontinence Sexual Questionnaire - validated measure for evaluation of sexuality
PFDI | One year
  Pelvic Floor Distress Inventory - validated measure for assessment of pelvic floor function
de novo stress urinary incontinence | One year
  complaints of the patient
de novo symptoms of overactive bladder | One year
  complaints of the patient
number of re-operations | One year
  for any reason
de novo dyspareunia | One year
  in previously sexually active women

CONTACTS AND LOCATIONS:
Overall Officials: Jaromir Masata, MD, Ph.D., Study Chair — Charles University, Czech Republic
Locations (2):
- Czechia (2):
  - General University Hospital, Prague, Prague
  - Vladimir Kalis, Pilsen